CLINICAL TRIAL: NCT03615261
Title: Promoting Healthy Brain Development Via Prenatal Stress Reduction: An Innovative Precision Medicine Approach: An Intervention Feasibility and Acceptability Pilot
Brief Title: Wellness For 2: A Feasibility and Acceptability Pilot
Acronym: We2-P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Sheila Krogh-Jespersen, Assistant Director, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STU00205776B
Record Dates: First submitted 2018-07-23; First posted 2018-08-03 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-10

CONDITIONS: Pregnancy; Prenatal Stress
Keywords: prenatal maternal stress; mindfulness; stress reduction; health sensing; mhealth

STUDY DESIGN:
Intervention Model Description: All participants engaged in the Mothers & Babies Intervention while wearing a biosensor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mothers and Babies (Enhanced) (Experimental): The course is a manualized stress-reduction intervention with an integrated tech suite designed for timely detection and response to stress. Based on Cognitive-Behavioral Therapy & attachment theory, MB is divided into 3 sections: Pleasant Activities; Thoughts; Contact with Others. Each module has been enhanced with mindfulness as a strategy to help "center" participants and facilitate practice of skills. Participants receive skills training in each of the three sections as tools to improve and manage their mood. The MB course emphasizes developing & strengthening the bond with the baby. The technology enhancement includes wearing a BioStamp sensor, and text message-based extra intervention content. Participants get worksheets linked to the 12 sessions.
  Interventions: Behavioral: Mothers and Babies (Enhanced)

INTERVENTIONS:
Behavioral: Mothers and Babies (Enhanced) — The course is a manualized stress-reduction intervention with an integrated tech suite designed for timely detection and response to stress. Based on Cognitive-Behavioral Therapy & attachment theory, MB is divided into 3 sections: Pleasant Activities; Thoughts; Contact with Others. Each module has been enhanced with mindfulness as a strategy to help "center" participants and facilitate practice of skills. Participants receive skills training in each of the three sections as tools to improve and manage their mood. The MB course emphasizes developing & strengthening the bond with the baby. The technology enhancement includes wearing a BioStamp sensor, and text message-based extra intervention content. Participants get worksheets linked to the 12 sessions.

SUMMARY:
The investigators are studying strategies and tools that women can use to manage stress and wellness during pregnancy. The purpose of this project is to test a technology-enhanced version of a wellness intervention for women during their pregnancy (the Mothers and Babies course; MB). The technology that the investigators will test includes wearable heart rate sensors, smartphone text message surveys, and intervention materials delivered through text message.

DETAILED DESCRIPTION:
Perinatal "early life" stress (ELS) has significant consequences for mothers and their infants.(1-3) Prolonged prenatal stress places pregnant women at increased risk for depression, health risk behaviors, and poor overall health and quality of life. Likewise, fetal exposure to stress places infants at greater risk of neurodevelopmental disruptions.(4,5)

Prior clinical trials led by co-PI Darius Tandon have demonstrated that pregnant women, particularly those in low income environments, demonstrate positive health and parenting benefits as a result of receiving prenatal stress reduction interventions.(6-8) The stress-reduction intervention proposed in the overarching Promoting Healthy Brains Project (PHBP), the Mothers and Babies course (MB), is a scalable, manualized evidence-based cognitive-behavioral intervention that can be adapted to meet client needs (e.g., setting, dose, timing, modality) without compromising fidelity. However, as there is substantial heterogeneity in maternal responsiveness to prenatal stress-reduction interventions, MB in its current form may be too low-intensity to improve fetal outcomes. Although a few studies have examined impact of interventions like MB on developmental outcomes, the extant evidence base does not provide strong support for intervention effects. Further, state-of-the-art neurodevelopmental methods have not been employed to detect how manipulation of early exposure to stress may effect brain:behavior patterns in early life. Advancing this is the overarching goal of the PHBP.

A crucial component of the proposed work involves an enhanced version of the 12-session, one-on-one version of MB with 1) mindfulness training content; 2) inter-session text messages prompting skills reinforcement, self-monitoring, and homework reminders; 3) adaptive, real-time stress monitoring that will optimize the intervention by identifying the key point at which to deliver just-in-time stress intervention content to individual participants.

The investigators will ask pregnant women to wear a long-wearing, unobtrusive wireless ECG sensor (BioStamp Research Connect; BioStamp). BioStamp sensor data will be used to detect physiological responses to stress (i.e., heart rate variability; HRV) to build a system that can be used to trigger real-time stress reduction intervention. BioStamp, a lightweight, rechargeable, and easy to use wearable device is equipped to passively and continuously measure HRV and motion. Unlike traditional "wired" ECG monitors, BioStamp can be worn under typical daily-living conditions (e.g., sleeping, showering, physical activity), with only minimal obtrusion in daily life (e.g., re-charging, re-applying adhesive).

Led by PI Laurie Wakschlag, the overarching PBHP will harness multidisciplinary expertise from Northwestern's Institute for Innovations in Developmental Sciences (DevSci), Lurie Children's Hospital, Center for Community Health, McCormick School of Engineering, and Feinberg School of Medicine & Northwestern Medicine (Ob/Gyn, Preventive Medicine, Medical Social Sciences, and Pediatrics) to 1) adapt and pilot MB enhanced with mindfulness training content, and just-in-time feedback to participants regarding their in-the-moment stress responses, and 2) experimentally test the effects of the optimized intervention on maternal wellbeing pre- and postnatally, and postnatal neurodevelopmental health trajectories.

ELIGIBILITY:
Inclusion Criteria:

* 10-18 weeks gestation
* singleton pregnancy
* receiving prenatal care from a Northwestern University prenatal care clinic & planning to deliver at Northwestern Hospitals
* English-speaking
* must own a smartphone
* must be willing to receive text messages and respond to short online surveys using their smartphone
* must also agree to wear a wireless adhesive sensor daily
* must have WiFi internet access for the duration of their participation in the study

Exclusion Criteria:

* have known chronic medical or pregnancy complications that may place their infant at risk for neurological disorders (e.g., HIV; acute cytomegalovirus infection (CMV); toxoplasmosis; zika virus; Phenylketonuria (PKU); chromosomal anomalies; metabolic disorder; substance use disorders)
* have significant mental health disorders (e.g., schizophrenia, bipolar disorder, psychosis) which could interfere with study adherence
* unable to wear the BioStamp Sensor due to known skin sensitivity (e.g., allergy to adhesives or silicone), current skin irritation, or broken skin at the placement site
* pacemaker or other sensitive medical device
* unable to provide informed consent, complete MB sessions, or complete study assessments in English
* currently participating in another MB course at the time of recruitment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Usability/Wearability Feedback | At post-intervention (approx. week 13)
  Participants will also be asked to provide survey feedback regarding the sensor's usability and wearability, and responding to the Environmental Momentary Assessments (EMAs).
Intervention Acceptability | After each of the 12 MB sessions (approx. weekly during weeks 2-13)
  All participants will complete a brief intervention rating checklist after completing each MB module (3 total). Additional acceptability information will be ascertained during the exit interview and survey at the end of the intervention to assess participants' overall ratings of the MB course, whether they would recommend the intervention to similar women, and suggestions for intervention modifications.

SECONDARY OUTCOMES:
Intervention fidelity | After each of the 12 MB sessions (approx. weekly during weeks 2-13)
  MB intervention fidelity delivered by facilitators will be measured by collecting data on a) intervention session completion and b) fidelity of intervention implementation. Facilitators will completed an intervention Facilitator Fidelity Rating Form immediately at the end of each visit. The fidelity rating form will measure 1) How much of each topic was covered; 2) How well the participant understood each topic; 3) participant engagement in each topic; 4) Any challenges when discussing the topic.
Ecological Momentary Assessment Subjective Stress Ratings | Five times daily for approx. weeks 1-13, and one week per month afterward until birth
  In-field, self-report EMAs will measure participants' negative and positive emotion, stress, and other factors (e.g., health behaviors) that may influence sensor readings. These surveys, delivered via text message, contain 4 questions on a 5-pt Likertscale from 'not at all' to 'very much', one on a 7-pt Likert scale from 'not at all' to 'very much', six on a binary yes/no scale, six on a visual analog scale from 'not at all' to 'extremely', and four for elaboration.
Objective stress response | Continuously during the intervention (approx. weeks 2-13)
  Investigators will continuously collect raw ECG and accelerometer data from the BioStamp Sensor.
Perceived Stress (State Trait Anxiety Inventory) | Day 1, post-intervention (approx. week 13), 1 month prior to, and 1 month after delivery
  40 questions about stress and anxiety-related feelings on a 4-pt Likert scale from 'Almost Never' to 'Almost Always'.
Perceived Stress (Life events scale distress rating) | Day 1, post-intervention (approx. week 13), 1 month prior to, and 1 month after delivery
  28 questions about the undesirability/negativity of a variety of life events that could happen to the participant or someone close to them on a 4-pt Likert scale from 'Not at all' to 'Very much'.
Perceived Stress (Perceived stress scale) | Day 1, post-intervention (approx. week 13), 1 month prior to, and 1 month after delivery
  10 questions about emotions on a 5-pt Likert scale of 'Never' to 'Very Often'
Depression symptoms (behavioral activation depression scale) | Day 1, post-intervention (approx. week 13), 1 month prior to, and 1 month after delivery
  25 questions about depressive feelings and behaviors on a 7-pt Likert scale from 'Not at All' to 'Completely'
Perceived stress (Prenatal Distress Questionnaire) | Day 1, post-intervention (approx. week 13), 1 month prior to, and 1 month after delivery
  17 questions about feeling bothered, worried, or upset on a 3-pt Likert scale from 'Not at all' to 'Very much'; Three open-ended questions to elaborate.
Depression symptoms (PROMIS depression) | Day 1, post-intervention (approx. week 13), 1 month prior to, and 1 month after delivery
  28 questions about depression-related thoughts and feelings on a 5-pt Likert scale from 'Never' to Always'
Depression symptoms (negative mood regulation scale) | Day 1, post-intervention (approx. week 13), 1 month prior to, and 1 month after delivery
  30 questions about depression-related thoughts and feelings on a 5-pt Likert scale from 'Strong disagreement' to 'Strong agreement'.
Depression symptoms (MOS social support survey) | Day 1, post-intervention (approx. week 13), 1 month prior to, and 1 month after delivery
  19 questions on feelings of support from others on a 5-pt Likert scale from 'None of the time' to 'All of the time'.
Depression symptoms (Experiences Questionnaire) | Day 1, post-intervention (approx. week 13), 1 month prior to, and 1 month after delivery
  20 questions about thoughts and feelings on a 5-pt Likert scale from 'Never' to 'All the time'.
Depression symptoms (Edinburgh depression scale) | Day 1, post-intervention (approx. week 13), 1 month prior to, and 1 month after delivery
  10 questions about negative emotions on a 4-pt Likert scale from 'No/Never' to 'Yes/A lot'.
Depression symptoms (Prenatal Health Behavior Scale) | Day 1, post-intervention (approx. week 13), 1 month prior to, and 1 month after delivery
  24 questions about diet, exercise, and drug use on a 5-pt Likert scale from 'Never' to 'Very Often'
Intervention skills (five facet mindfulness questionnaire) | Day 1, post-intervention (approx. week 13), 1 month prior to, and 1 month after delivery
  39 questions about mindfulness behaviors on a 5-pt Likert scale from 'Never or very rarely true' to 'Very often or always true'
Intervention skills (MB skills use survey) | Day 1, post-intervention (approx. week 13), 1 month prior to, and 1 month after delivery
  35 questions about intervention skill use frequency (5-pt Likert scale from 'Every Day' to 'Not at all'), helpfulness and enjoyability (3-pt Likert scales from 'Not at all' to 'Very')

CONTACTS AND LOCATIONS:
Overall Officials: Lauren S Wakschlag, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Talge NM, Neal C, Glover V; Early Stress, Translational Research and Prevention Science Network: Fetal and Neonatal Experience on Child and Adolescent Mental Health. Antenatal maternal stress and long-term effects on child neurodevelopment: how and why? J Child Psychol Psychiatry. 2007 Mar-Apr;48(3-4):245-61. doi: 10.1111/j.1469-7610.2006.01714.x. PMID 17355398
- [Background] Kinsella MT, Monk C. Impact of maternal stress, depression and anxiety on fetal neurobehavioral development. Clin Obstet Gynecol. 2009 Sep;52(3):425-40. doi: 10.1097/GRF.0b013e3181b52df1. PMID 19661759
- [Background] O'Connor TG, Heron J, Golding J, Glover V; ALSPAC Study Team. Maternal antenatal anxiety and behavioural/emotional problems in children: a test of a programming hypothesis. J Child Psychol Psychiatry. 2003 Oct;44(7):1025-36. doi: 10.1111/1469-7610.00187. PMID 14531585
- [Background] de Bruijn AT, van Bakel HJ, van Baar AL. Sex differences in the relation between prenatal maternal emotional complaints and child outcome. Early Hum Dev. 2009 May;85(5):319-24. doi: 10.1016/j.earlhumdev.2008.12.009. Epub 2009 Jan 21. PMID 19162414
- [Background] Grizenko N, Fortier ME, Zadorozny C, Thakur G, Schmitz N, Duval R, Joober R. Maternal Stress during Pregnancy, ADHD Symptomatology in Children and Genotype: Gene-Environment Interaction. J Can Acad Child Adolesc Psychiatry. 2012 Feb;21(1):9-15. PMID 22299010
- [Background] Mendelson T, Leis JA, Perry DF, Stuart EA, Tandon SD. Impact of a preventive intervention for perinatal depression on mood regulation, social support, and coping. Arch Womens Ment Health. 2013 Jun;16(3):211-8. doi: 10.1007/s00737-013-0332-4. Epub 2013 Mar 2. PMID 23456540
- [Background] Tandon SD, Leis JA, Mendelson T, Perry DF, Kemp K. Six-month outcomes from a randomized controlled trial to prevent perinatal depression in low-income home visiting clients. Matern Child Health J. 2014 May;18(4):873-81. doi: 10.1007/s10995-013-1313-y. PMID 23793487
- [Background] Tandon SD, Perry DF, Mendelson T, Kemp K, Leis JA. Preventing perinatal depression in low-income home visiting clients: a randomized controlled trial. J Consult Clin Psychol. 2011 Oct;79(5):707-12. doi: 10.1037/a0024895. PMID 21806298